CLINICAL TRIAL: NCT01538771
Title: The Efficacy of IntraCoronary Erythropoietin Delivery BEfore Reperfusion: Gauging Infarct Size in Patients With Acute ST-segment Elevation Myocardial Infarction (ICEBERG).
Brief Title: Intracoronary Darbepoetin-alpha to Reduce The Infarct Size and Post-Infarct Remodeling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAMI
Record Dates: First submitted 2012-02-15; First posted 2012-02-24 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Erythropoietin; Myocardial reperfusion injury
MeSH Terms: conditions — Myocardial Infarction; Myocardial Reperfusion Injury | interventions — Darbepoetin alfa; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): Received same volume of saline
  Interventions: Drug: Control Saline
- Darbepoetin group (Active Comparator): Darbepoetin alfa 300ug intracoronary bolus infusion via over-the-wire balloon before the 1st ballooning & conventional treatment
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoetin alfa 300ug intracoronary bolus infusion via over-the-wire balloon before the 1st ballooning and conventional treatment
  Other Names: Nesp PFS Prefilled Syringe (Jeilkirin Pharm. Korea)
  Arms: Darbepoetin group
Drug: Control Saline — Same volume of saline intracoronary bolus infusion via over-the-wire balloon before the 1st ballooning and conventional treatment
  Other Names: 0.9% normal saline
  Arms: Control group

SUMMARY:
Prospective, randomized and open label trial

Hypothesis

* Infusion of intracoronary darbepoetin-alpha at the time of reperfusion may reduce infarct size and post-infarct pathologic left ventricular remodeling in patients with ST-segment elevation myocardial infarction.

Methods

* Randomization into control group or treatment group
* Treatment group : Darbepoetin-alpha 300ug intracoronary bolus infusion via over-the-wire balloon system simultaneously with first balloon inflation and conventional treatment
* Control group : conventional treatment

Endpoints

* peak CK-MB & troponin levels : baseline,6h,12hr,18hr, 24hr, 36hr and 48hr
* MRI at baseline : infarct size, area at risk and salvaged myocardium
* MRI at 4 months : prevalence of pathologic left ventricle remodeling (definition: increase of end-diastolic volume index > 20% compared to baseline)
* safety endpoint : cardiac death, nonfatal myocardial infarction, stent thrombosis, ischemic stroke, hospital readmission with heart failure or ischemic symptom, bleeding and urgent target lesion revascularization

DETAILED DESCRIPTION:
[Eligibility Criteria]

1. Patients, regardless of gender, at the age from 18 to 80 years were eligible if they had within 12 hours of onset of ST-segment myocardial infarction that was decided to treat with primary percutaneous coronary intervention.

[Exclusion criteria]

1. Uncontrolled congestive heart failure (Killip classes II and III, or cardiogenic shock)
2. History of malignancy
3. Serious hematological disease
4. Current infectious disease requiring antibiotic therapy
5. Baseline creatinine level > 2.0 mg/dL or dependence on dialysis
6. Known hypersensitivity to or contraindication for heparin, aspirin, clopidogrel, sirolimus, everolimus, contrast medium and darbepoetin-α

[Primary endpoint] Myocardial infarct size, estimated by measurement of peak levels of cardiac biomarker (CK-MB and troponin-I of the patients was followed for 48 hours at every 6 hours)

[Secondary end points]

1. The infarct size, measured as the area of delayed enhancement seen with cardiac magnetic resonance (CMR) imaging on average four days after ST-segment elevation myocardial infarction (baseline)
2. The proportion of area at risk (AAR) and salvaged myocardium, calculated by formula; [AAR - Infarct size] / AAR X 100 (%)
3. The change of left ventricular ejection fraction (LVEF), LV end-diastolic volume (LVEDV), and LV end-systolic volume (LVESV) assessed by CMR between four days and four months
4. LV remodeling index [(LVEDV at four months - baseline LVEDV) / baseline LVEDV X 100%] and the incidence of pathologic LV remodeling (LV remodeling index > 20%);

[Safety endpoints] The incidence of composites of the cardiovascular endpoints (cardiac death, nonfatal myocardial infarction, stent thrombosis, ischemic stroke, hospital readmission with heart failure or ischemic symptoms, bleeding and urgent target lesion revascularization) assessed at four months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-elevation myocardial infarction (MI) within 12 hours of onset
* Suitable coronary anatomy for PCI
* Age < 80 yrs

Exclusion Criteria:

* Uncontrolled congestive heart failure (Killip classes II and III, or cardiogenic shock)
* History of malignancy
* Serious hematological disease
* Current infectious disease requiring antibiotic therapy
* Baseline creatinine level > 2.0 mg/dL or dependence on dialysis
* Known hypersensitivity to or contraindication for heparin, aspirin, clopidogrel, sirolimus, everolimus, contrast medium and darbepoetin-α

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Peak CK-MB/ Troponin-I levels | baseline, 6, 12,18,24,36,48hrs

SECONDARY OUTCOMES:
Infarct size, area at risk and proportion of salvaged myocardium | Participants will be followed for the duration of hospital stay, an expected average of 4 days
  Assessed by cardiac MRI
Pathologic left ventricle remodeling assessed by cardiac MRI | 4 months
  Definition : Increase of end-diastolic volume of left ventricle >20%
Change of left ventricular ejection fraction, LV end-diastolic volume , and LV end-systolic volume assessed by cardiac MRI | Between four days and 4 months
Composites of cardiovascular endpoints | 4 Months
  ccardiac death, nonfatal myocardial infarction, stent thrombosis, ischemic stroke, hospital readmission with heart failure or ischemic symptoms, bleeding and target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Suh JW, Yoon YE, Oh IY, Yoon CH, Cho YS, Youn TJ, Chae IH, Choi DJ. A single-center prospective randomized controlled trial evaluating the safety and efficacy of IntraCoronary Erythropoietin delivery BEfore Reperfusion: gauging infarct size in patients with acute ST-segment elevation myocardial infarction. Study design and rationale of the 'ICEBERG Trial'. Contemp Clin Trials. 2013 May;35(1):145-50. doi: 10.1016/j.cct.2013.03.001. Epub 2013 Mar 16. PMID 23506972